CLINICAL TRIAL: NCT02125292
Title: A Phase 1, Open-label, Randomized, 3-period Crossover Taste Assessment Study to Characterize the Palatability of SHP429 When the Contents Are Sprinkled Onto Soft Foods or Emptied Into a Cup and Administered With Water in Healthy Adult Subjects
Brief Title: Taste Assessment Study of SHP429 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SHP429-102
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — Mesalamine

ARMS (3):
- Mesalamine (Vanilla Yogurt) (Experimental): One 500mg capsule contents sprinkled onto 1 tablespoon of low-fat vanilla yogurt
  Interventions: Drug: Mesalamine
- Mesalamine (Applesauce) (Experimental): One 500mg capsule contents sprinkled onto 1 tablespoon of applesauce
  Interventions: Drug: Mesalamine
- Mesalamine (Dosing Cup) (Experimental): One 500mg capsule contents emptied into a dosing cup and taken with water
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: Mesalamine
  Other Names: Pentasa, SHP429

SUMMARY:
The purpose of this study is to compare the palatability of SHP429 capsule contents delivered via 3 means of administration (sprinkled on yogurt, sprinkled on applesauce, and emptied into a cup and administered with water).

ELIGIBILITY:
Inclusion Criteria:

* normal, healthy, adult male and female volunteers, without evidence of active or chronic disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2014-06-19 (Actual); Study Completion 2014-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesalamine in Vanilla Yogurt, Then Applesauce, Then Water; Mesalamine in Applesauce, Then Water, Then Vanilla Yogurt; Mesalamine in Applesauce, Then Vanilla Yogurt, Then Water; Mesalamine in Vanilla Yogurt, Then Water, Then Applesauce; Mesalamine in Water, Then Vanilla Yogurt, Then Applesauce; Mesalamine in Water, Then Applesauce, Then Vanilla Yogurt: Three different modes of administration were tested. Treatment A: 1 SHP429 500mg capsule opened and the contents sprinkled onto 1 tablespoon of commercially available low-fat vanilla yogurt and the contents were then administered to the participant; Treatment B: 1 SHP429 500mg capsule opened and the contents sprinkled onto 1 tablespoon of commercially available unsweetened, creamy applesauce and the contents were then administered to the participant; Treatment C: 1 SHP429 500mg capsule opened and the contents emptied into a dosing cup, the contents were then administered to the participant. The participant was administered 240mL of room temperature water to aid in the consumption of the capsule content.
Period: First Intervention (1 Hour)
Arm/Group | Mesalamine in Vanilla Yogurt, Then Applesauce, Then Water | Mesalamine in Applesauce, Then Water, Then Vanilla Yogurt | Mesalamine in Applesauce, Then Vanilla Yogurt, Then Water | Mesalamine in Vanilla Yogurt, Then Water, Then Applesauce | Mesalamine in Water, Then Vanilla Yogurt, Then Applesauce | Mesalamine in Water, Then Applesauce, Then Vanilla Yogurt
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (2 Hours)
Arm/Group | Mesalamine in Vanilla Yogurt, Then Applesauce, Then Water | Mesalamine in Applesauce, Then Water, Then Vanilla Yogurt | Mesalamine in Applesauce, Then Vanilla Yogurt, Then Water | Mesalamine in Vanilla Yogurt, Then Water, Then Applesauce | Mesalamine in Water, Then Vanilla Yogurt, Then Applesauce | Mesalamine in Water, Then Applesauce, Then Vanilla Yogurt
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Hour)
Arm/Group | Mesalamine in Vanilla Yogurt, Then Applesauce, Then Water | Mesalamine in Applesauce, Then Water, Then Vanilla Yogurt | Mesalamine in Applesauce, Then Vanilla Yogurt, Then Water | Mesalamine in Vanilla Yogurt, Then Water, Then Applesauce | Mesalamine in Water, Then Vanilla Yogurt, Then Applesauce | Mesalamine in Water, Then Applesauce, Then Vanilla Yogurt
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (2 Hours)
Arm/Group | Mesalamine in Vanilla Yogurt, Then Applesauce, Then Water | Mesalamine in Applesauce, Then Water, Then Vanilla Yogurt | Mesalamine in Applesauce, Then Vanilla Yogurt, Then Water | Mesalamine in Vanilla Yogurt, Then Water, Then Applesauce | Mesalamine in Water, Then Vanilla Yogurt, Then Applesauce | Mesalamine in Water, Then Applesauce, Then Vanilla Yogurt
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Hour)
Arm/Group | Mesalamine in Vanilla Yogurt, Then Applesauce, Then Water | Mesalamine in Applesauce, Then Water, Then Vanilla Yogurt | Mesalamine in Applesauce, Then Vanilla Yogurt, Then Water | Mesalamine in Vanilla Yogurt, Then Water, Then Applesauce | Mesalamine in Water, Then Vanilla Yogurt, Then Applesauce | Mesalamine in Water, Then Applesauce, Then Vanilla Yogurt
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race [Count of Participants; unit: Participants]
  White | 16
  Non-white, black or African American | 2
Weight [Mean (Standard Deviation); unit: kilograms] | 67.59 (13.312)
Height [Mean (Standard Deviation); unit: centimeters] | 166.2 (9.25)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.348 (3.4331)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Responses to Palatability Assessment of The Taste of Mesalamine
Description: A taste assessment was completed immediately after investigational product was administered to assess the subject's taste/liking of the formulation. The assessment consisted of a 5-point rating scale. Participants were asked to choose one of the following responses to the statement "The taste was acceptable": strongly agree, agree, neutral, disagree, or strongly disagree. The number of participants who chose either of the top two responses (strongly agree, agree) is reported.
Time Frame: Immediately post-dose
Population: Pharmacodynamic Set: all participants who took at least 1 dose of investigational product and had at least 1 post-dose taste assessment.
Measure: Number; unit: participants
Groups:
- Mesalamine (Vanilla Yogurt): One 500mg Mesalamine capsule opened and the contents sprinkled onto 1 tablespoon of commercially available low-fat vanilla yogurt. All 3 treatments were administered on the same day, with a 2-hour washout period between investigational product administrations in each treatment period.
- Mesalamine (Applesauce): One 500mg Mesalamine capsule opened and the contents sprinkled onto 1 tablespoon of commercially available unsweetened, creamy applesauce. All 3 treatments were administered on the same day, with a 2-hour washout period between investigational product administrations in each treatment period.
- Mesalamine (Dosing Cup): One 500mg Mesalamine capsule opened and the contents emptied into a dosing cup; contents were then administered to the subject with 240ml of water. All 3 treatments were administered on the same day, with a 2-hour washout period between investigational product administrations in each treatment period.
Arm/Group | Mesalamine (Vanilla Yogurt) | Mesalamine (Applesauce) | Mesalamine (Dosing Cup)
Number analyzed (Participants) | 18 | 18 | 18
participants | 17 | 16 | 13

2. Primary Outcome: Number of Participants Who Detected an Aftertaste of Mesalamine
Description: An aftertaste assessment was completed 5 minutes after administration of investigational product to assess whether the participants detected an aftertaste. The participants answered "Yes" or "No" to the following question: "Was there an aftertaste?" The number of participants who answered "Yes" is reported.
Time Frame: 5 minutes post-dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Mesalamine (Vanilla Yogurt) | Mesalamine (Applesauce) | Mesalamine (Dosing Cup)
Number analyzed (Participants) | 18 | 18 | 18
participants | 0 | 4 | 1

3. Primary Outcome: Number of Participants With Positive Responses to Palatability Assessment of The Aftertaste of Mesalamine
Description: An aftertaste assessment was completed 5 minutes after administration of investigational product to assess the subject's rating of aftertaste and means of administration. The assessment consisted of a 5-point rating scale. The participants were asked to choose one of the following responses to the statement "The aftertaste (if present) was acceptable": strongly agree, agree, neutral, disagree, or strongly disagree. The number of participants who chose either of the top two responses (strongly agree, agree) is reported.
Time Frame: 5 minutes post-dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Mesalamine (Vanilla Yogurt) | Mesalamine (Applesauce) | Mesalamine (Dosing Cup)
Number analyzed (Participants) | 18 | 18 | 18
participants | 0 | 3 | 1

4. Primary Outcome: Number of Participants Willing to Take Mesalamine Via Treatment Method on a Regular Basis
Description: The participants were asked to answer "Yes" or "No" to the following question: "Would you be willing to take medicine this way on a regular basis if necessary?" The number of participants who answered "Yes" is reported.
Time Frame: Immediately post-dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Mesalamine (Vanilla Yogurt) | Mesalamine (Applesauce) | Mesalamine (Dosing Cup)
Number analyzed (Participants) | 18 | 18 | 18
participants | 18 | 17 | 18

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event
Description: Participants were monitored for treatment-emergent adverse events through the follow-up assessment, which occurred 2 days +/- 1 day post-dose.
Time Frame: 4 days
Population: Safety Set: all participants who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Number; unit: participants
Groups:
- All Participants: All participants who received all 3 treatments
Arm/Group | All Participants
Number analyzed (Participants) | 18
participants
  Serious Adverse Event | 0
  Non-serious Adverse Event | 2

6. Secondary Outcome: Number of Participants With Potentially Clinically Important Laboratory Results
Description: Clinical laboratory assessments included hematology, chemistry and urinalysis parameters, all measured 6 hours post-dose. All clinical laboratory assays were performed according to the laboratory's normal procedures. Reference ranges were supplied by the laboratory and were used to assess the clinical laboratory data for clinical significance and out-of-range pathological changes. The investigator assessed out-of-range clinical laboratory values for clinical significance and indicated whether or not the values were clinically significant.
Time Frame: 1 day
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 18
participants
  Hematology | 0
  Biochemistry | 0
  Urinalysis | 3

7. Secondary Outcome: Number of Participants With Potentially Clinically Important Vital Signs
Description: Vital sign assessments included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate and body temperature measurements, all measured 6 hours post-dose. Study personnel used both absolute values and change from baseline values to determine if the vital sign was potentially clinically important. Criteria for the potential clinical importance of both absolute and change from baseline values were pre-specified. A participant's vital sign had to meet both the absolute and change from baseline criteria to be considered as potentially clinically important.
Time Frame: 1 day
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 18
participants | 0

8. Secondary Outcome: Number of Participants With Potentially Clinically Important Electrocardiogram (ECG) Results
Description: Subjects underwent a standard 12-lead ECG 6 hours post-dose. The investigator assessed if the ECG tracing was normal or abnormal; if abnormal, the investigator made a determination of whether or not the abnormality was clinically significant.
Time Frame: 1 day
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 18
participants | 0

ADVERSE EVENTS:
Time Frame: 4 days
Arm/Group | Mesalamine (Vanilla Yogurt) | Mesalamine (Applesauce) | Mesalamine (Dosing Cup)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 1/18 | 0/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalamine (Vanilla Yogurt) (N=18) | Mesalamine (Applesauce) (N=18) | Mesalamine (Dosing Cup) (N=18)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.